CLINICAL TRIAL: NCT01775826
Title: Validating Machine -Learned Classifiers of Sedentary Behavior and Physical Activity
Acronym: iWatch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Marta Jankowska, Prinicipal Investigator, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1R01CA164993-01A1 (NIH)
Record Dates: First submitted 2013-01-17; First posted 2013-01-25 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Physical Activity; Sedentary Lifestyle
Keywords: physical activity; sedentary behavior; accelerometer; GPS; GIS; machine learning
MeSH Terms: conditions — Motor Activity; Sedentary Behavior | interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Purposes (Other): All participants.
  Interventions: Other: Measurement

INTERVENTIONS:
Other: Measurement — Measured usual (day-to-day) behavior with body-worn sensors.

SUMMARY:
The majority of the US population spends most of the day sitting and the we have new scientific evidence that this can contribute to poor health regardless of how much physical activity a person does. However, we do not measure sitting time very accurately and when we ask people to tell us how much they do, their answers are unreliable. Our study will use small sensors to objectively measure when people sit or do physical activity, and we will use sophisticated computational techniques to summarize these movement patterns.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for participants 6-17 yr olds:

* provide written parental consent to complete study protocols;
* provide verbal assent to complete study protocols;
* willingness to complete 2 visits to UCSD offices;
* willingness to wear multiple sensor devices on 7 days for 12 hours per day;
* willingness to wear wrist accelerometer on 7 days for 24 hours per day;
* willingness to have their height and weight measured;
* be able to walk unassisted
* able to read and understand study materials in English.

Inclusion Criteria for participants 18-64 yr old:

* provide written consent to complete study protocols;
* willingness to complete 2 visits to UCSD offices;
* willingness to wear multiple sensor devices on 7 days for 12 hours per day;
* willingness to wear wrist accelerometer on 7 days for 24 hours per day;
* complete a survey assessing their demographic characteristics;
* willingness to have their height and weight measured;
* be physically and cognitively able to walk unassisted,
* able to read and understand study materials in English.

Inclusion Criteria for participants 65-85 yr olds:

* provide written consent to complete study protocols;
* correctly answer verbal questions about their comprehension of the informed consent;
* willingness to complete 2 visits to UCSD offices;
* willingness to wear multiple sensor devices on 7 days for 12 hours per day;
* willingness to wear wrist accelerometer on 7 days for 24 hours per day;
* complete a survey assessing their demographic;
* willingness to have their height and weight measured;
* be physically and cognitively able to walk without the assistance of another person (walking aids are permitted)
* able to read and understand study materials in English.

Exclusion Criteria:

* unable to ambulate;
* attends a workplace or school on monitoring days that prohibits static images being taken by a SenseCam worn around the neck of the participant;
* pregnancy in second or third trimester.

Ages: 6 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2013-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
physical activity behavior classification using study sensors (accelerometers, Sensecam and GPS) | Baseline
  Using an annotated data set of SenseCam images in three free-living population subgroups, we will compare sensitivity, specificity and percent agreement between behavioral classifiers derived from: (a) single axis vs. multi axis accelerometers; (b) aggregated movement counts vs. raw acceleration data; (c) hip vs. wrist mounted accelerometers.
  Determine (a) the extent to which adding GPS data improves discrimination accuracy over accelerometer only behavior classification (i.e., best classifier resulting from Aim 1); and (b) the extent to which adding GIS data improves discrimination accuracy over accelerometer and GPS behavior classification alone (i.e., best classifier resulting from Aim 2a).

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD, La Jolla, California, United States

REFERENCES:
- [Background] Moghimi, Mohammad**; Kerr, Jacqueline; Johnson, Eileen; Godbole, Suneeta; Belongie, Serge Discriminative Regions: A Substrate for Analyzing Life-Logging Image Sequences MultiMedia Modeling 2015 357-368.
- [Background] Kerr J, Patterson RE, Ellis K, Godbole S, Johnson E, Lanckriet G, Staudenmayer J. Objective Assessment of Physical Activity: Classifiers for Public Health. Med Sci Sports Exerc. 2016 May;48(5):951-7. doi: 10.1249/MSS.0000000000000841. PMID 27089222
- [Background] Ellis K, Kerr J, Godbole S, Staudenmayer J, Lanckriet G. Hip and Wrist Accelerometer Algorithms for Free-Living Behavior Classification. Med Sci Sports Exerc. 2016 May;48(5):933-40. doi: 10.1249/MSS.0000000000000840. PMID 26673126